## Official title: Impact of exercise on expression of Hsp70 in individuals at risk of peripheral arterial disease.

NCT ID: Not yet assigned

Document's date: December 11, 2020

| CONTROL GROUP | | | | | EXPERIMENTAL GROUP | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Data<br>median, SD<br>and mean | Median at the beginning | Median at the end | Difference<br>beginning -<br>end | p | Data median,<br>SD and mean | Median at the beginning | Median at the end | Difference<br>beginning -<br>end | p |
| Weight (kg) | $67.35 \pm 11.99$ | $66.44 \pm 11.76$ | -0.91 | 0.008* | Weight (kg) | $70.00 \pm 11.94$ | $69.88 \pm 12.66$ | -0.12 | 0.587 |
| | 66.45 | 65.9 | -0.55 | | | 67 | 67.9 | 0.9 | |
| BMI<br>(Kg/m²) | $27.73 \pm 4.68$ | $27.73 \pm 4.60$ | 0 | 0.066 | BMI (Kg/m²) | $28.85 \pm 3.26$ | 29.21 ± 3.97 | 0.36 | 0.364 |
| | 27.35 | 28.6 | -1.75 | | | 27.7 | 28.25 | 0.55 | |
| WC (cm) | $90.18 \pm 9.76$ | 89.53 ± 10.55 | -0.65 | 0.394 | WC (cm) | 92.42±11.38 | 90.53 ±13.37 | -1.89 | 0.629 |
| | 90.6 | 89.5 | -1.1 | | | 89 | 90.5 | 1.5 | |
| WHtR | $0.58 \pm 0.06$ | $0.57 \pm 0.06$ | 0 | 0.363 | WHtR | 0.59 ±0.06 | 0.58 ±0.07 | 0 | 0.756 |
| | 0.59 | 0.59 | 0 | | | 0.59 | 0.6 | 0.01 | |
| ABI<br>(mmHg) | $0.95 \pm 0.02$ | $0.98 \pm 0.11$ | 0.04 | 0.147 | ABI (mmHg) | 0.95 ±0.02 | 1.00 ±0.05 | 0.05 | 0.001* |
| | 0.95 | 0.99 | 0.04 | | | 0.95 | 0.99 | 0.04 | |
| Systolic BP (mmHg) | 128.12 ± 18.83 | 120 ± 15.00 | -8.12 | 0.069 | Systolic BP (mmHg) | 124 ±19.93 | 118.43 ±12.38 | -5.57 | 0.209 |
| | 130 | 120 | -10 | | | 117.5 | 118 | 0.5 | |
| Diastolic BP<br>(mmHg) | $79.18 \pm 14.29$ | $73.62 \pm 8.02$ | -5.56 | 0.059 | Diastolic BP<br>(mmHg) | 76.37±10.13 | 73.31 ±8.86 | -3.06 | 0.080 |
| | 80 | 73.62 | -6.38 | | | 74 | 73.5 | -0.5 | |
| RHR (bpm) | $78.25 \pm 11.61$ | $73.43 \pm 13.19$ | -4.82 | 0.14 | RHR (bpm) | 78.31 ±13.34 | 62.75 ±8.53 | -15.56 | 0.00* |
| | 76.5 | 71.5 | -5 | | | 80 | 61.5 | -18.5 | |
| Sit and reach | $10.40 \pm 12.09$ | $11.12 \pm 10.51$ | 0.72 | 0.706 | Sit and reach | 10.25 ±7.75 | $9.71 \pm 8.32$ | -0.54 | 0.779 |
| | 8.25 | 13.75 | 5.5 | | | 8 | 9 | 1 | |
| Hsp 70<br>(pg/mL) | 0.04 ±0.0 | 0.04 ±0.0 | 0 | 0.004* | Hsp 70<br>(pg/mL) | 0.04 ±0.00 | 0.03 ±0.00 | -0.01 | 0.005* |
| | 0.04 | 0.04 | 0 | | | 0.04 | 0.03 | -0.01 | |

\*W de Mann (Wilcoxon) test, significant p Value in bold Body Mass Index: BMI, Waist Circumference: WC, Ankle-Brachial Index: ABI, Blood Pressure: BP, Resting Heart Rate: RHR.